CLINICAL TRIAL: NCT03454074
Title: B-Fit Intervention to Improve Engagement in Healthy Brain Aging Activities in Middle-aged and Older Adults
Brief Title: B-Fit Intervention to Improve Brain Health
Acronym: B-Fit
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Washington State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: WashingtonSU
Record Dates: First submitted 2016-02-15; First posted 2018-03-05 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Health Behavior; Aging
Keywords: healthy aging; behavior change; older adults
MeSH Terms: conditions — Health Behavior | interventions — Educational Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- B-Fit intervention (Experimental): Combines group education about brain health with individualized goal-setting and group problem-solving to help participants effectively integrate healthy behavioral changes into their everyday lives.
  Interventions: Behavioral: Problem-solving; Behavioral: Education
- Education Only (Active Comparator): Provide group education about healthy behavior changes without problem-solving component.
  Interventions: Behavioral: Education
- Wait-list (No Intervention): No intervention administered. Will be offered intervention following a delay.

INTERVENTIONS:
Behavioral: Problem-solving — Individualized goal-setting and group problem-solving to help older adults effectively integrate realistic, healthy behavioral changes into their everyday lives
  Arms: B-Fit intervention
Behavioral: Education — Education about healthy brain aging behaviors provided.
  Arms: B-Fit intervention; Education Only

SUMMARY:
An accumulating body of research indicates that activities such as exercise, active cognitive and social engagement, good sleep hygiene, stress reduction and proper nutrition are associated with the maintenance of cognitive health. Emerging data also suggests that healthy lifestyle behaviors may promote brain plasticity. Despite nationwide efforts to raise public awareness about brain health, there remains a gap concerning how to best promote behavioral change and help at-risk middle-aged and older adults adopt effective, evidence-based brain health behaviors into their everyday lives to maximize cognitive health. The objective of this study is to evaluate the efficacy of a 7-week group brain fitness intervention (B-Fit) for increasing preventative brain health behaviors and enhancing cognitive health in participants at-risk for cognitive impairment. We will also examine mechanisms of action of the B-Fit intervention through tracking of behavioral responses in the real-world environment using wearable sensors.

DETAILED DESCRIPTION:
Participants will be middle-aged and older adults. Participants will be randomized to one of three conditions (B-fit, education only, wait-list). Outcome measures will be administered at baseline, post-treatment and at a one-year follow-up. Participants will also be asked to wear an actigraph for 7 days at baseline, post intervention and follow-up. One or two clinicians will lead the intervention groups, which will each have 8-12 group members. Both the B-Fit and education control conditions will meet 2 hours per week for 7 weeks. Participants in both conditions will receive identical educational materials provided in the form of weekly learning packets and presented to the group by the study clinician(s). At the first meeting, group members will be presented with an overview of the brain, cognitive aging, mild cognitive impairment, and dementia. Each subsequent group meeting will cover a specific topic. The topics will be presented to all groups in the following order: cognitive engagement, exercise and cardiovascular risk factors, nutrition, social engagement, sleep and stress reduction, and compensatory strategy use. The control condition will include presentation of the educational materials followed by expanded discussion about the materials among group members. In contrast, each meeting of the B-Fit intervention will follow a highly structured format. The format is designed to aid participants in identifying and setting realistic and valuable individualized brain health goals and in obtaining group support through problem-solving, modeling and encouragement.

ELIGIBILITY:
Inclusion Criteria:

* Age 40+ (midlife and older adults)

Exclusion Criteria:

* Adults under the age of 40
* Adults who meet criteria for dementia
* Adults who cannot provide own informed consent
* Adults who cannot complete assessments or participate in the intervention protocols due to vision, hearing, communication or other difficulties
* Adults unable to read and comprehend information in English.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-02-15 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Healthy Aging Activity Engagement | Change in engagement in healthy brain aging behaviors as measured by the HAAE from baseline to post-test (appr. 2 months) and follow-up (appr. one-year).
  (Subjective Measure) Healthy Aging Activity Engagement Scale (HAAE): participants use a 5-point Likert scale to rate level of agreement with engagement in healthy brain behaviors during the past week from strongly disagree (0) to strongly agree (5). Scores range from 32 to 160, with higher scores representing greater engagement in positive health behaviors.
Objective sensor-based behavior change detection with wearable sensors | Change in activities captured by actigraphs and measured using a behavior change detection approach at baseline compared to post-test (appr. 2 months) and follow-up (appr. one-year).
  (Objective Measure) Participants will wear an Actigraph for 1 week to capture objective data in the form of activity times, activity durations, mobility, activity level and sleep/time quality. We will apply the behavior change detection approach (BCD) to detect the magnitude of health-related changes in behavior patterns and to describe the nature of the changes (e.g., increased afternoon activity).

SECONDARY OUTCOMES:
Physical Capability | Change in mobility as measured by the SPPB from baseline to post-test (appr. 2 months) and follow-up (appr. one-year).
  The Short Physical Performance Battery (SPPB) will provide a composite measure of physical capability. The SPPB combines the results of gait speed, chair stand and balance tests.
Psychological Wellbeing | Change in psychological wellbeing as measured by the total score of the NIH Toolbox surveys from baseline to post-test (appr. 2 months) and follow-up (appr. one-year).
  The concept of psychological well-being will be captured by the NIH Toolbox surveys that measure the following three components: positive affect, general life satisfaction, and meaning and purpose. A total score will be computed.
Cognitive Function | Change in fluid cognitive abilities as measured by the NIH Toolbox fluid cognition composite from baseline to post-test (appr. 2 months) and follow-up (appr. one-year).
  NIH Toolbox Fluid Cognition Composite Score will be used to assess for change in cognition.
Social Wellbeing | Change in social wellbeing as measured by the total score of the NIH surveys from baseline to post-test (appr. 2 months) and follow-up (appr. one-year).
  The concept of social wellbeing will be captured by by the NIH Toolbox surveys that measure the following components: emotional support, friendship, instrumental support, loneliness, perceived hostility, and perceived rejection. A total score will be computed.

CONTACTS AND LOCATIONS:
Overall Officials: Maureen Schmitter-Edgecombe, Ph.D., Principal Investigator — Washington State University
Locations (1):
- Washington State University, Pullman, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Boyd B, McAlister C, Arrotta K, Schmitter-Edgecombe M. Self-Reported Behavior Change and Predictors of Engagement With a Multidomain Brain Health Intervention for Midlife and Older Adults: A Pilot Clinical Trial. J Aging Health. 2022 Jan;34(1):109-119. doi: 10.1177/08982643211032483. Epub 2021 Jul 15. PMID 34266343